CLINICAL TRIAL: NCT00002387
Title: A Multicenter, Open, Randomized, Forty-Eight-Week, Pilot Study to Evaluate the Activity, Safety, and Pharmacokinetics of Indinavir Sulfate, 1200 Mg q 12h and DMP 266, 300 Mg q 12h Versus Indinavir Sulfate, 1000 Mg q 8h and DMP 266, 600 Mg q.h.s.
Brief Title: The Safety and Effectiveness of Indinavir Sulfate Plus Efavirenz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 246K; 067-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Drug Administration Schedule; HIV Protease Inhibitors; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; efavirenz
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Indinavir; efavirenz

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Efavirenz

SUMMARY:
To estimate the differences in parameters of antiviral activity and safety between a control regimen of indinavir in combination with DMP 266 and an experimental regimen of higher-dose indinavir in combination with lower-dose DMP 266 after sixteen weeks of dosing, in protease inhibitor- and non-nucleoside reverse transcriptase inhibitor-naive, HIV-1 seropositive patients.

It is hypothesized that after 16 weeks of randomized treatment with either the control or experimental regimen that:

1. The observed proportion of patients with serum viral RNA < 400 copies/ml in the experimental and control regimen will be similar and will continue to be so after 48 weeks.
2. The safety profiles of the two groups will be similar, judged by the incidence of serious, drug-related adverse experiences and the incidence of events of specific interest (e.g., nephrolithiasis, hyperbilirubinemia, nausea/vomiting, rash, and CNS-related symptoms) and will continue to be so after 48 weeks.
3. The two groups will be similar with respect to changes from baseline in serum viral RNA and CD4 counts and will continue to be so after 48 weeks.

DETAILED DESCRIPTION:
It is hypothesized that after 16 weeks of randomized treatment with either the control or experimental regimen that:

1. The observed proportion of patients with serum viral RNA < 400 copies/ml in the experimental and control regimen will be similar and will continue to be so after 48 weeks.
2. The safety profiles of the two groups will be similar, judged by the incidence of serious, drug-related adverse experiences and the incidence of events of specific interest (e.g., nephrolithiasis, hyperbilirubinemia, nausea/vomiting, rash, and CNS-related symptoms) and will continue to be so after 48 weeks.
3. The two groups will be similar with respect to changes from baseline in serum viral RNA and CD4 counts and will continue to be so after 48 weeks.

Patients are randomized to one of two regimens: a control regimen of indinavir plus DMP 266 or an experimental regimen of indinavir plus DMP 266, each at different doses than in the control regimen.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositive status.
* CD4 count >= 100 cells/mm3.
* Serum viral RNA levels >= 10,000 copies/ml.

Exclusion Criteria

Prior Medication:

Excluded:

* Prior protease inhibitor therapy.
* Prior non-nucleoside reverse transcriptase inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCSD Treatment Ctr / Dept of Medicine & Pediatrics, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - Hawaii AIDS Clinical Trial Unit, Honolulu, Hawaii
  - Rush Med Ctr / Section of Infectious Diseases, Chicago, Illinois
  - Beth Israel Hosp, Boston, Massachusetts
  - Univ Hosp / SUNY at Stony Brook / AIDS TMT Unit, Stony Brook, New York
  - Brown Univ / Miriam Hosp, Providence, Rhode Island